CLINICAL TRIAL: NCT04165824
Title: Safety Study of Oral Edaravone Administered in Subjects With ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1186-A01
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Results first posted 2022-08-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ALS
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT-1186 (Experimental)
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — * An initial treatment cycle with daily dosing for 14 days, followed by a 14-day drug free period
  * Subsequent treatment cycles with daily dosing for 10 days out of a 14-day period, followed by a 14 day drug free period. Treatment cycles are every 4 weeks.
  Other Names: Oral edaravone

SUMMARY:
The objective of this study is to evaluate the long-term safety and tolerability of oral edaravone in subjects with Amyotrophic Lateral Sclerosis (ALS) over 24 and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female, ≥ 18 to 75 years of age at the time the ICF is signed
* Subjects will be diagnosed with Definite ALS, Probable ALS, Probable laboratory-supported ALS, or Possible ALS according to the El Escorial revised criteria for the diagnosis of ALS.
* Subjects will be living and functioning independently (eg, able to eat, excrete, ambulate independently without assistance of others). The use of supportive tools and adaptive utensil is allowed
* Subjects will have a baseline forced vital capacity percentage (%FVC) ≥ 70%.
* Subjects whose first symptom of ALS occurred within 3 years of the time of providing written informed consent.

Exclusion Criteria:

* Subjects who have the presence or history of any clinically significant disease (except ALS) that could interfere with the objectives of the study (the assessment of safety and efficacy) or the safety of the subject, as judged by the Investigator.
* Subjects of childbearing potential unwilling to use acceptable method of contraception from the screening visit until 3 months after the last dose of study medication. Subjects who are sexually active who do not agree to use contraception during the study period.
* Subjects who are female and pregnant (a positive pregnancy test) or lactating at the screening visit (Visit 1).
* Subjects who have a significant risk of suicidality. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the 3 months before the screening visit.
* Subjects who have ALT or AST elevations greater than 2 times the ULN at screening.
* Subjects with a Glomerular Filtration Rate (GFR) <30 mL/Min Per 1.73 m2.
* Subjects with history of hypersensitivity to edaravone, any of the additives or inactive ingredients of edaravone, or sulfites.
* Subjects with hereditary fructose intolerance.
* Subjects who participated in another study and were administered an investigational product within 1 month or 5 half-lives of the investigational agent, whichever is longer before providing informed consent for the present study.
* Subjects who are unable to take their medications orally.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science,, Study Director — Tanabe Pharma America, Inc.
Locations (53):
- United States (22):
  - St. Joseph's Hospital and Medical Center (SJHMC) - Barrow Neurological Institute (BNI) - The Gregory W. Fulton ALS and Neuromuscular Disease Center, Phoenix, Arizona
  - Neuromuscular Research Center, Phoenix, Arizona
  - Woodland Research Northwest, Rogers, Arkansas
  - Sutter Health, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UF Health Cancer Center, Gainesville, Florida
  - Emory University - School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan - ALS Center of Excellence, Ann Arbor, Michigan
  - University of Michigan Health System (UMHS) - Allergy Clinic - Northville Health Center Location, Northville, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Neurology Associates, P.C - Lincoln, Lincoln, Nebraska
  - Wake Forest University Baptist Medical Center (WFUBMC) - The J. Paul Sticht Center on Aging and Rehabilitation, Winston-Salem, North Carolina
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - Wesley Neurology Clinic, P.C., Cordova, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - UT Health Science Center San Antonio, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Heritage Medical Research Clinic - University Of Calgary, Calgary, Alberta
  - University of Alberta - Walter C Mackenzie Health Sciences Centre (WCM), Edmonton, Alberta
  - Recherche Sepmus, Inc, Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (5):
  - CHU Nice-Hospital Archet I, Nice, Alpes Maritimes
  - Centre Hospitalier Esquirol, Limoges, Marcland
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Hopital Pierre Wertheimer - Hopital Neurologique, Bron
  - CHU de NICE Hopital Pasteur 2 -Centre de Reference des Maladies -Neuromusculaires & SLA-Pole Neurosciences Cliniques, Nice
- Germany (2):
  - Deutsche Klinik fuer Diagnostik, Wiesbaden, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Italy (3):
  - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan, MI
  - Universita degli Studi di Torino - Centro Regionale Esperto Per La Sclerosi Laterale Amiotrofica (CRESLA), Turin, Piedmont
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca Granda - Centro Clinico Nemo (Neuro Muscular Omnicentre), Milan
- Japan (17):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - National Hospital Organization Chiba-East-Hospital, Chiba, Chiba
  - Murakami Karindoh Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - National Hospital Organization Iou National Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Kumamoto Saishun Medical Center, Koshi-shi, Kumamoto
  - National Hospital Organization Utano Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical And Dental Hospital, Niigata, Niigata
  - National Hospital Organization Toneyama Medical Center, Toyonaka-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Genge A, Pattee GL, Sobue G, Aoki M, Yoshino H, Couratier P, Lunetta C, Petri S, Selness D, Bidani S, Hirai M, Sakata T, Salah A, Apple S, Wamil A, Kalin A, Jackson CE. Oral edaravone demonstrated a favorable safety profile in patients with amyotrophic lateral sclerosis after 48 weeks of treatment. Muscle Nerve. 2023 Feb;67(2):124-129. doi: 10.1002/mus.27768. Epub 2022 Dec 28. PMID 36504406

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-1186: MT-1186 105mg (2 weeks On/Off)
Period: Overall Study
Arm/Group | MT-1186
Started | 185
Completed | 139
Not Completed | 46
Not completed — Adverse Event | 23
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 17
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | MT-1186
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.9)
Age, Customized [Count of Participants; unit: Participants]
  20 to 29 years | 1
  30 to 39 years | 6
  40 to 49 years | 19
  50 to 59 years | 60
  60 to 69 years | 63
  >=70 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 177
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergency Adverse Events
Time Frame: up to 48 Weeks
Measure: Number; unit: events
Arm/Group | MT-1186
Number analyzed (Participants) | 185
events | 961

2. Primary Outcome: Number of Participants With Treatment Emergency Adverse Events
Time Frame: Up to 48 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MT-1186
Number analyzed (Participants) | 185
Participants | 175

3. Other Pre Specified Outcome: Change in ALS Functional Rating Scale - Revised From Baseline
Time Frame: up to 48 Weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Time to Event (Death, Tracheostomy, and Permanent Assisted Mechanical Ventilation)
Time Frame: up to 48 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 48 weeks
Arm/Group | MT-1186
All-Cause Mortality (participants affected / at risk) | 12/185
Serious Adverse Events (participants affected / at risk) | 48/185
Other Adverse Events (participants affected / at risk) | 123/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=185)
Cellulitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Feeding disorder (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 12
Muscle spasticity (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 6
Pelvic pain (Reproductive system and breast disorders) | 1
Gait disturbance (General disorders) | 1
Pain (General disorders) | 1
Oxygen saturation decreased (Investigations) | 1
Weight decreased (Investigations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Patella fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Gastrostomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=185)
Constipation (Gastrointestinal disorders) | 33
Dysphagia (Gastrointestinal disorders) | 16
Salivary hypersecretion (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 14
Contusion (Injury, poisoning and procedural complications) | 15
Fall (Injury, poisoning and procedural complications) | 40
Back pain (Musculoskeletal and connective tissue disorders) | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Muscular weakness (Musculoskeletal and connective tissue disorders) | 39
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 13
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT04165824/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT04165824/SAP_001.pdf